CLINICAL TRIAL: NCT05554016
Title: The UFO (Ultra Processed Foods in Obesity) Project
Acronym: UFO Project
Status: Recruiting | Type: Observational
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Professor of Pediatrics, Federico II University
Other Study IDs: 00019173
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Obesity, Morbid; Metabolic Syndrome
MeSH Terms: conditions — Obesity, Morbid; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group 1: Pediatric patients with obesity
- Group 2: Pediatric patients with obesity complicated by Metabolic Syndrome
- Group 3: Age- and sex-matched healthy controls

SUMMARY:
The childhood obesity prevalence has increased dramatically in the last decades, affecting more than 340 million children worldwide. This condition is the major risk factor for a set of metabolic abnormalities, also known as metabolic syndrome, a condition that reduce life expectancy by 5-20 years. Changes in the global food system, and the increased consumption of ultra-processed foods (UPFs), may have contributed to the increase in the prevalence of childhood obesity and related morbidities. The mechanisms by which UPFs might promote obesity and metabolic syndrome could be multiple and not completely identified.

The Ultra-processed Food in Obesity (UFO) Project has been designed to investigate the potential associations between UPFs intake and MetS in pediatric subjects

ELIGIBILITY:
Inclusion Criteria:

* Caucasian ethnicity, both sexes, age ≥6 and ≤18 years, diagnosis of obesity (Group 1), diagnosis of obesity and Metabolic Syndrome (Group 2), and age- and sex-matched healthy controls (Group 3).

Exclusion Criteria:

* Non-Caucasian ethnicity;
* Age <6 or >18 years;
* Concomitant presence of chronic diseases, neoplasms, immunodeficiencies, chronic infections,autoimmune diseases, chronic inflammatory bowel disease, celiac disease, metabolic-genetic diseases, cystic fibrosis and other chronic lung diseases, cardiovascular/respiratory/gastrointestinal malformations, neuropsychiatric disorders, and neurological disorders;
* Intake of antibiotics and/or pre/pro/synbiotics;
* History of obesity surgery and onset of diarrhea or acute gastrointestinal illness during the 12 weeks prior to enrollment;
* Presence of tattoos, scars, moles or special lesions on both forearms.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric subjects of caucasian ethnicity, of both sexes, aged ≥6 and ≤18 years, with a sure diagnosis of obesity (Group 1), of obesity complicated by Metabolic Syndrome (Group 2), and age- and sex-matched healthy controls (Group 3).
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Dietary UPF intake | At enrollment
  The assessment of dietary UPF intake will be carried out through a 7-day food diary.

SECONDARY OUTCOMES:
Daily intake of energy and nutrients | At enrollment
  The daily intake of energy (kcal) and nutrients will be carried out through a 7-day food diary.
Daily dietary intake of AGEs | At enrollment
  The intake of Advanced Glycation Endproducts (mostly present in UPFs).
Skin AGEs levels | At enrollment
  The skin accumulation of AGEs in the subcutaneous.
RAGE expression in peripheral blood mononuclear cells | At enrollment
  The expressione of the AGEs receptor in peripheral blood mononuclear cells.
Soluble form of RAGE expression | At enrollment
  The expressione of the AGEs receptor in the serum.
Mitochondrial metabolism | At enrollment
  The mitochondrial metabolism through the Seahorse XFp analyzer.
Oxidative stress | At enrollment
  Oxidative stress biomarkers.
Interleukin-6 | At enrollment
  Serum levels of Interleukin-6.
MicroRNA-221 expression | At enrollment
  MicroRNA-221 expression in peripheral blood mononuclear cells.
Leptin | At enrollment
  Serum levels of leptin.
Ghrelin | At enrollment
  Serum levels of ghrelin.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Traslational Medical Science - University of Naples Federico II, Naples, Italy

IPD SHARING:
Plan to Share IPD: No